CLINICAL TRIAL: NCT05942300
Title: Phase I Trial of CPI-0209 in Combination With Carboplatin in Patients With Platinum Sensitive Recurrent Ovarian Cancer
Brief Title: CPI-0209 Plus Carboplatin in Patients With Platinum Sensitive Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lan Coffman (Other)
Collaborators: Novartis Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lan Coffman, Hematology/Oncology. Assistant Professor of Medicine., University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-249; CA272218 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Ovarian Cancer
Keywords: platinum sensitive; stromal tumor microenvironment (TME); PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-0209 (100 mg) + carboplatin (Experimental): CPI-0209: 100 mg (oral dosing) carboplatin administered intravenously as per institutional standards
  Interventions: Drug: CPI-0209; Drug: carboplatin
- CPI-0209 (150 mg) + carboplatin (Experimental): CPI-0209: 100 mg (oral dosing) carboplatin administered intravenously as per institutional standards
  Interventions: Drug: CPI-0209; Drug: carboplatin

INTERVENTIONS:
Drug: CPI-0209 — A second-generation EZH2 inhibitor that has been designed to achieve comprehensive anti-cancer target coverage through extended on-target residence time.
  Other Names: Tulmimetostat
Drug: carboplatin — Carboplatin is a chemotherapy drug that contains the metal platinum. It stops or slows the growth of cancer cells and other rapidly growing cells by damaging their DNA.

SUMMARY:
This is a clinical trial using CPI-0209 in combination with Carboplatin chemotherapy followed by CPI-0209 maintenance in patients with platinum sensitive, recurrent ovarian cancer.

DETAILED DESCRIPTION:
Clinically, there is a critical need for improved therapies in ovarian cancer. There has been recent success with maintenance therapy in ovarian cancer with both PARP inhibitors and bevacizumab approved in the up-front maintenance setting and in the recurrent, platinum sensitive maintenance setting. However, it is unclear what treatment should be used post-PARPi or bevacizumab maintenance. Additionally, the benefit derived from bevacizumab maintenance therapy is modest with generally a few month improvement in progression free survival. Further, there is emerging evidence that after progression on a PARPi, there is decreased response to platinum-based therapy. This provides a critical unmet need to enhance platinum response, particularly after previous maintenance therapy. This also provides a large group of patients who could potentially benefit from EZH2 targeting agents to block stromal-mediated chemotherapy resistance and metastasis.

This study aims to investigate whether CPI-0209 will enhance ovarian cancer sensitivity to platinum-based chemotherapy and prolong the disease free interval after completion of chemotherapy by blocking stromal mediated chemotherapy resistance, metastasis promotion and ovarian cancer growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with platinum-sensitive recurrent ovarian, fallopian or primary peritoneal cancer (defined as recurrent disease > 6 months after completing last platinum- based chemotherapy) that are eligible to receive platinum-based chemotherapy).
* Documented disease recurrence/progression based on GCIG-RECIST
* Must have had at least 1 prior line of platinum-based therapy, prior bevacizumab or PARPi use are allowed. Women with germline BRCA mutations should be considered for PARPi maintenance as standard of care treatment prior to consideration of clinical trial enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 with life expectancy of ≥ 3months
* Adequate organ function

  * Serum creatinine ≤1.5mg/dL or 24-hour clearance ≥50mL/min
  * AST/ALT <2.5x ULN (or <5x ULN if liver metastasis are present)
  * Total bilirubin ≤ ULN or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome
  * Hemoglobin ≥9 gm/dl, Platelets ≥100,000/μl ANC ≥1500/μl
  * INR ≤1.5
  * Potassium, total calcium (corrected for serum albumin), magnesium, and sodium within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
* Must be able to swallow CPI-0209 tablet/oral suspension
* Able to provide informed consent and comply with all study protocol
* Treated CNS metastasis allowed if treatment is completed ≥8 weeks prior to enrollment. Patients must be asymptomatic off systemic corticosteroids for at least 4 weeks after completion of radiation therapy. CNS disease must be stable or regressed on repeat imaging performed at least 4 weeks after completion of therapy.
* Women of child-bearing potential (those who have had a menstrual cycle within the last year and have not had a tubal ligation or surgical removal of both ovaries and/or hysterectomy) must agree to abstain from vaginal intercourse or use and continue highly effective methods of contraception for at least 183 days after discontinuation of study treatment.

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient.
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Exclusion Criteria:

* Borderline or low malignant potential histology
* Platinum-resistant disease (as defined as progressive disease (PD) within 6 months of completion of chemotherapy with a platinum agent).
* Known hypersensitivity to any of the excipients of CPI-0209.
* Gastrointestinal (GI) dysfunction or disease that may significantly alter the absorption of the study drugs
* Concurrent malignancy or malignancy within 3 years prior to starting study drug with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer or per physician discretion that the previous cancer was adequately treated with curative intent and unlikely to recur (the study PI must concur with this determination).
* History of HIV infection
* Has an active infection requiring systemic treatment
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks and contraindicate patient's participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, significant cardiac/pulmonary disease etc.)
* Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Use of herbal supplements unless discontinued ≥7 days prior to initiation of study drug
* Consumption of foods which are strong inducers or inhibitors of CYP3A4/5 has to be discontinued 7 days prior to initiation of study drug. Patients that are unwilling to exclude Seville oranges, grapefruit juice, AND grapefruit from the diet and all foods that contain those fruits from time of enrollment to through the duration of study participation will be excluded.
* Pregnant or breast feeding
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
* Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated.
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 5 Grade ≤1 (Exception to this criterion: patients with any grade of alopecia, controlled endocrine toxicities and/or neuropathy ≤ grade 2 are allowed to enter the study).
* Grade 3 baseline neuropathy
* Patient with a Child-Pugh score B or C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of CPI-0209 | Up to 24 months
  MTD will be determined via Dose-limiting toxicity (DLT)s defined as any grade 3-4 non-hematological or grade 4 hematological toxicity at least possibly related to the treatment, occurring during the first two cycles of treatment and per Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Adverse Events by Grade per CTCAE v5.0 | Up to 5.5 years
  Number of patients that experienced grade 3 or greater Adverse events per the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 5, determined to be at least possibly, probably or definitely related to treatment.
Overall Response Rate (ORR) | 5.5 years
  Proportion of patients with Complete Response (CR) or Partial Response (PR) per RECIST v 1.1. Per RECIST v1.1: CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. PR is defined as ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free Survival (PFS) | Up to 5.5 years
  The length of time during and after treatment that a patient lives with disease but without disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Coffman, MD, PhD, Principal Investigator — UPMC Magee Women's Hospital
Locations (1):
- Magee-Womens Research Institute / UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No